CLINICAL TRIAL: NCT01055132
Title: Dispensing Evaluation of New Daily Disposable Toric Soft Contact Lens.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1476AG
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etafilcon A toric contact lens/Nelfilcon A toric (Other): Etafilcon A toric contact lens first, then nelfilcon A toric second
  Interventions: Device: Etafilcon A toric contact lens; Device: Nelfilcon A toric contact lens
- Nelfilcon A toric/ Etafilcon A toric (Other): Nelfilcon A toric contact lens first, then etafilcon A toric toric second
  Interventions: Device: Etafilcon A toric contact lens; Device: Nelfilcon A toric contact lens

INTERVENTIONS:
Device: Etafilcon A toric contact lens — contact lens to correct astigmatism
Device: Nelfilcon A toric contact lens — contact lens to correct astigmatism

SUMMARY:
The purpose of this study is to determine the relative performance of a new daily disposable toric soft contact lens against a daily disposable toric contact lens currently available in market, specifically with regards to the comfort and vision with the lens.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be between 18 and 40 years old.
* The subject must have normal eyes.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must read and sign the STATEMENT OF INFORMED CONSENT and be provided a copy of the form.
* The subject must have a subjective distance spectacle prescription in the range of -1.75 to -5.00D in each eye.
* The subject must manifest -1.25 to -2.00 D of refractive astigmatism in each eye.
* The subject's refractive cylinder axis must be 180 degrees plus or minus 30 degrees in each eye.
* The subject must be an adapted wearer of soft toric contact lenses in both eyes.
* The subject's best visual acuity (BVA) must be better than or equal to 20/25 in each eye.
* Subjects must already possess a wearable pair of spectacles.

Exclusion Criteria:

* Ocular or systemic allergies or disease that may interfere with contact lens wear.
* Systemic disease or autoimmune disease or use of medication, which may interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining or any other abnormality of the cornea, which may contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities that might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation
* Any infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* Diabetes
* Strabismus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Los Angeles, California
  - Jacksonville, Florida
  - Marietta, Georgia
  - New York, New York
  - Warwick, Rhode Island

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject failed screening, and did not enter group assignment
Groups:
- Etafilcon A Toric Lens First/ Nelfilcon A Toric Lens Second: Etafilcon A toric contact lens worn daily during first period of 5 - 9 days, then nelfilcon A toric contact lens worn daily during second period of 5 - 9 days
- Nelfilcon A Toric Lens First/Etafilcon A Toric Lens Second: Nelfilcon A toric contact lens worn daily during first period of 5 - 9 days, then etafilcon A toric contact lens worn daily during second period of 5 - 9 days
Period: Period 1 (5-9 Days)
Arm/Group | Etafilcon A Toric Lens First/ Nelfilcon A Toric Lens Second | Nelfilcon A Toric Lens First/Etafilcon A Toric Lens Second
Started | 36 | 33
Completed | 35 | 33
Not Completed | 1 | 0
Not completed — unsatisfactory lens fitting performance | 1 | 0
Period: Period 2 (5-9 Days)
Arm/Group | Etafilcon A Toric Lens First/ Nelfilcon A Toric Lens Second | Nelfilcon A Toric Lens First/Etafilcon A Toric Lens Second
Started | 35 | 33
Completed | 35 | 32
Not Completed | 0 | 1
Not completed — Unsatisfactory lens fitting performance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who completed the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Monocular Visual Acuity on LogMAR Scale
Description: Distance (4 meter) high contrast standard resolution (ETDRS) acuity was measured twice for each eye. Visual acuity describes the acuteness or sharpness of vision; the ability to perceive small details. Visual acuity is a measure of spacial resolution of the visual processing system; it's tested by requiring the person being tested to identify characters (like letters and numbers)on a chart from a set distance. LogMAR charts are used to assess visual acuity for research studies. LogMAR means Minimum Angle of Resolution. This has lead to the assertion that research is done using a logarithmic progression in size of letters on a test chart gives the most accurate visual acuity measurement. The reason for this is, unlike other charts, LogMAR chart has equal gradation between the letters on the line and the space between the lines. And, there is a fixed number of letters per line.
Time Frame: After 5 to 9 days of lens wear
Population: Analysis was conducted on subjects who successfully complete the study.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Etafilcon A Toric (Test Lens): Etafilcon A toric is a daily disposable hydrogel toric lens with the addition of a wetting agent, developed for a wider ranged of prescriptions; worn for 5-9 days
- Nelfilcon A Toric (Active Comparator): An existing, daily disposable toric contact lens; worn 5-9 days
Arm/Group | Etafilcon A Toric (Test Lens) | Nelfilcon A Toric (Active Comparator)
Number analyzed (Participants) | 67 | 67
logMAR | -0.065 (0.0777) | -0.038 (0.1057)
Statistical Analysis 1: Comparison: Etafilcon A Toric (Test Lens) vs Nelfilcon A Toric (Active Comparator); Ho:The test lens is non-inferior to the active comparator lens for monocular visual performance on logMAR scale at 1-week follow-up. A non-inferiority margin of 0.05 logMAR was used; Test type: Non-Inferiority or Equivalence — Based on historical data, a minimum of 42 subjects is needed to achieve 80% power with 0.05 type I error; linear mixed model; Sequence of wear, period and lens were included as fixed effects; site, patient, eye*patient, period*patient and period*eye*patient as random effects; Least-square mean difference = -0.037, 95% CI 2-sided [-0.041 to -0.0013], Standard Error of Mean 0.0072 — Comparison between study lenses was carried out using 2-sided 95% confidence interval of the least-square mean difference(test minus control). The non-inferiority was concluded if the upper limit of the confidence limit is below 0.05 LogMAR

2. Primary Outcome: Binocular Visual Acuity on LogMAR Scale
Description: Distance (4 meter) high contrast standard resolution (ETDRS) acuity was measured twice binocularly. Distance (4 meter) high contrast standard resolution (ETDRS) acuity was measured twice for each eye. Visual acuity describes the acuteness or sharpness of vision; the ability to perceive small details. Visual acuity is a measure of spacial resolution of the visual processing system; it's tested by requiring the person being tested to identify characters (like letters and numbers)on a chart from a set distance. LogMAR charts are used to assess visual acuity for research studies. LogMAR means Minimum Angle of Resolution. This has lead to the assertion that research is done using a logarithmic progression in size of letters on a test chart gives the most accurate visual acuity measurement. The reason for this is, unlike other charts, LogMAR chart has equal gradation between the letters on the line and the space between the lines. And, there is a fixed number of letters per line.
Time Frame: After 5 to 9 days of lens wear
Population: Analysis was conducted on subjects who successfully complete the study.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Nelfilcon A Toric Lens (Active Comparator): An existing, daily disposable toric contact lens; worn 5-9 days
Arm/Group | Etafilcon A Toric (Test Lens) | Nelfilcon A Toric Lens (Active Comparator)
Number analyzed (Participants) | 67 | 67
LogMAR | -0.122 (0.0718) | -0.108 (0.0766)
Statistical Analysis 1: Comparison: Etafilcon A Toric (Test Lens) vs Nelfilcon A Toric Lens (Active Comparator); Ho:The test lens is non-inferior to the active comparator lens for Binocular visual performance on logMAR scale at 1-week follow-up. A non-inferiority margin of 0.05 logMAR was used; Test type: Non-Inferiority or Equivalence — Based on historical data, a minimum of 42 subjects is needed to achieve a minimum of 80% power with 0.05 type I error; linear mixed model; Sequence of wear,lens period and lens were included in the model as fixed effects; site, patient, period*patient were included as random effects; Least-square mean difference = -0.015, 95% CI 2-sided [-0.027 to -0.003], Standard Error of Mean 0.0062 — Comparison between study lenses was carried out using 2-sided 95% confidence interval of the least-square mean difference (test minus control). The non-inferiority was concluded if the upper limit of the confidence limit is below 0.05 LogMAR

3. Primary Outcome: Subject Reported Overall Lens Comfort Using the Contact Lens User Evaluation (CLUE)TM Questionnaire
Description: The Contact Lens User Evaluation(CLUE)TM questionnaire is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3*SD).
Time Frame: After 5 to 9 days of lens wear
Population: Analysis was conducted on subjects who successfully complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A (Test Lens): Etafilcon A toric is a daily disposable hydrogel toric lens with the addition of a wetting agent, developed for a wider ranged of prescriptions; worn 5-9 days
- Nelfilcon A (Active Comparator): An existing, daily disposable toric contact lens; worn for 5-9 days
Arm/Group | Etafilcon A (Test Lens) | Nelfilcon A (Active Comparator)
Number analyzed (Participants) | 67 | 67
units on a scale | 56.4 (9.12) | 44.0 (9.34)
Statistical Analysis 1: Comparison: Etafilcon A (Test Lens) vs Nelfilcon A (Active Comparator); Ho:The test lens is non-inferior to the active comparator lens for comfort at 1-week follow-up. A non-inferiority margin of -5 units was used; Test type: Non-Inferiority or Equivalence — Based on historical data, a minimum of 42 subjects is needed to achieve a minimum of 80% power with 0.05 type I error; linear mixed model; Sequence of lens wear, lens period and lens type were included in the model as fixed effects; and Site and patient as random effects; Least-square mean difference = 11.9, 95% CI 2-sided [4.05 to 19.79], Standard Error of Mean 3.93 — Comparison between study lenses was carried out using 2-sided 95% confidence interval of the least-square mean difference (test minus control). The non-inferiority was concluded if the lower limit of the confidence interval is higher than -5

4. Primary Outcome: Subject Reported Overall Quality of Vision Using the Contact Lens User Evaluation(CLUE)TM Questionnaire.
Description: as for outcome 3
Time Frame: After 5 to 9 days of lens wear
Population: Analysis was conducted on subjects who successfully complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A (Test Lens): Etafilcon A toric is a daily disposable hydrogel toric lens with the addition of a wetting agent, developed for a wider ranged of prescriptions; worn for 5-9 days
Arm/Group | Etafilcon A (Test Lens) | Nelfilcon A (Active Comparator)
Number analyzed (Participants) | 67 | 67
units on a scale | 52.7 (8.64) | 44.7 (9.41)
Statistical Analysis 1: Comparison: Etafilcon A (Test Lens) vs Nelfilcon A (Active Comparator); Ho:The test lens is non-inferior to the active comparator lens for overall quality of vision at 1-week follow-up. A non-inferiority margin of -5 units was used; Test type: Non-Inferiority or Equivalence — Based on historical data, a minimum of 42 subjects is needed to achieve a minimum of 80% power with 0.05 type I error; linear mixed model; [statistical method as in outcome 3, analysis 1]; least-square mean difference = 7.7, 95% CI 2-sided [0.58 to 14.80], Standard Error of Mean 3.55 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Groups:
- Etafilcon A Toric / Nelfilcon A Toric: etafilcon A toric contact lens worn daily during first period of a maximum of 9 days, nelfilcon A toric contact lens worn during second period of a maximum of 9 days
Arm/Group | Etafilcon A Toric / Nelfilcon A Toric
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications require agreement and written approval from Sponsor.